CLINICAL TRIAL: NCT01764139
Title: Vitamin D Levels In Patients Who Has Normal to Grade 2 Knee Arthroscopy Changes or Who Did Not Improve Symptoms Following Minor Knee Arthroscopic Procedures
Brief Title: Vitamin D Levels In Patients Who Has Normal to Grade 2 Knee Arthroscopy Changes
Status: Terminated | Type: Observational
Why Stopped: Lack of patients with recruitment criteria
Sponsor: Dr. S R Thanthulage (Other)
Responsible Party: Sponsor-Investigator, Dr. S R Thanthulage, DR, Mid Essex Hospital NHS Trust
Organization: Mid Essex Hospital NHS Trust (Other)
Other Study IDs: 12/LO/1689; 12/LO/1689 (Other: Directory of NRES Research Ethics Committees)
Record Dates: First submitted 2013-01-07; First posted 2013-01-09 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Knee Pain
Keywords: Minimal knee changes
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Knee pain patients with minimal knee changes: Male & no pregnant female age between 18-40 yrs.
  Interventions: Procedure: Blood sampling

INTERVENTIONS:
Procedure: Blood sampling
  Other Names: Investigtion of Vitamin D levels

SUMMARY:
Vitamin D deficiency has long been linked to musculoskeletal pain, and many other chronic disease conditions. Vitamin D is a nutrient that functions as a hormone precursor, and wide-ranging health effects are supported by the presence of vitamin D receptors in several cell types and tissues of the body (eg, lymphocytes and monocytes, brain, heart, pancreas, intestine, and placenta).In addition to its essential role of maintaining bone health, hypovitaminosis D has been implicated in the development of serious conditions, including diabetes, various types of cancer, and cardiovascular diseases.

Vitamin D is a unique prohormone that humans obtain in small amount from food, dietary supplements and largely by endogenous skin synthesis from 7-dehydrocholesterol with sunlight exposure. This endogenous synthesis produces the form vitamin D3 (cholecalciferol).Vitamin D deficiency and insufficiency are very common in the UK. Local audit at Chelmsford has shown severe deficiency of vitamin D among chronic pain patients.

The major source of vitamin D synthesis relies on sunlight exposure which is likely to be affected by modern lifestyles, which increasingly involve working indoors during daylight hours. This may be particularly important when combined with residence in northern latitudes and a cloudy climate.The proposed pilot study aims to identify percentage of vitamin D deficiency among knee pain patients by investigating eligible patients' blood for '25 hydroxy vitamin D'.

English speaking patients whose knee pain has not been resolved following knee arthroscopy are eligible for the study. Study will be carried out at the Broomfield hospital chronic pain department.

Duration will be around 6 months.

DETAILED DESCRIPTION:
Introduction Vitamin D deficiency has recently been linked with a range of diseases including chronic pain. Range of vitamin D levels are classified as deficiency less than 50nmols, insufficient 50 to 75 nmols, and adequate 75 to 150 nmoles, excessive more than 150nmol. Vitamin D deficiency was also identified in some of the chronic pain patients who presented to our pain clinic at Broomfield hospital.

Vitamin D deficiency and insufficiency are very common in the UK. Local audit at Chelmsford has shown severe deficiency of vitamin D among chronic pain patients.

The major source of vitamin D synthesis relies on sunlight exposure which is likely to be affected by modern lifestyles, or increasingly working indoors during daylight hours. This may be particularly important when combined with residence in northern latitudes and a cloudy climate.

Observational and circumstantial evidence suggests that there may be a role for vitamin D treatment for some chronic pain conditions. Al-Jarallah &colleagues had showed that (25(OH) D level was 11.4 ± 6.07 ng/ml.) 92.9% were vitamin D deficient among their Kuwaiti patients with primary knee osteoarthritis (21).

Our aim is to identify how many percentages of our patients, who are having knee pain, without any major abnormal findings are deficient of vitamin D.

If this number is significant, can we supplement them to improve their pain? If we correctly supplement patients early enough, can we prevent further deterioration of their knee joint? These are some of the questions we may be able to investigate and treat.

Currently the investigations of vitamin D levels were done on patients with primary knee osteoarthritis and to assess its relation with radiological grading and functional status, but not to assess the relationship with pain.

Research Aims, hypotheses We aim to identify incidence of vitamin D deficiency among knee pain patients. If this proves significant, next step is to organise a trial to treat these patients to identify the effectiveness of adequate supplementation for relieving pain. Our aim is to investigate around 50 patients.

Recruitment English speaking patients whose knee pain has not been resolved following knee arthroscopy will be invited to the study. Sample size will be only 50 patients. Patients will explain the purpose of the study in plain English before the invitation. After giving informed consent, sample of blood will be taken for '25hydroxy vitamin D' levels. Study will be carried out at the Broomfield hospital chronic pain department.

Inclusion criteria Male & no pregnant female age between 18-40 yrs, who continue to experience knee pain following normal to Grade 2 knee arthroscopy findings.

Exclusion Criteria Any types of anatomical or neurological causes for the pain, history of seizures, regional pain syndrome, alcohol or drug abuse, and malignancy, patients with clinically significant diseases and patients who do not understand English will be excluded.

Intervention or procedure One blood sample per patient.

Data management and analysis The proportion of patients with vitamin D deficiency will be estimated from the data and the corresponding 95% confidence limits calculated using the Wilson method. The mean and standard deviation of the vitamin D level will be estimated from the data along with the corresponding 95% confidence limits obtained using a bootstrap with 999 samples. The statistical distribution of the vitamin D level will also be examined.

Primary outcome measure for the study To identify the percentages of Vitamin D deficiency among the knee pain patients

ELIGIBILITY:
Inclusion Criteria:

* Male & no pregnant female age between 18-40 yrs, who continue to experience knee pain following normal to Grade 2 knee arthroscopy findings.

Exclusion Criteria:

* Any types of anatomical or neurological causes for the pain, history of seizures, regional pain syndrome, alcohol or drug abuse, and malignancy, patients with clinically significant diseases and patients who do not understand English will be excluded.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Male & no pregnant female age between 18-40 yrs, who continue to experience knee pain following normal to Grade 2 knee arthroscopy findings.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2013-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
The percentages of Vitamin D deficiency among the knee pain patients. | 6months
  To identify the percentages of Vitamin D deficiency among the knee pain patients

CONTACTS AND LOCATIONS:
Locations (1):
- Broomfield Hospital, Chelmsford, Essex, United Kingdom